CLINICAL TRIAL: NCT00985764
Title: Venous Air Embolism in Cesarean Delivery, Especially Placental Previa
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Ki Jun Kim, Yonsei University, College of Medicine, Dep of Anesthesiology
Other Study IDs: 4-2007-0006
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-10

CONDITIONS: Cesarean Delivery With Placental Previa
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- placental previa
  Interventions: Procedure: cesarean delivery

INTERVENTIONS:
Procedure: cesarean delivery

SUMMARY:
Effects of placenta previa on incidence and severity of venous air embolism in patients during cesarean delivery

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer with cesarean delivery

Exclusion Criteria:

* the one who rejects to participate

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: cesarean delivery with placental previa
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
read sonography records during the surgery | After 1 or 2 weeks of surgery
  Three sono views will be recorded rapidly for later interpretation of the stage of air embolism. The midesophageal (ME) 4-chamber view will be continuously monitored during surgery and videotaped. When a bubble is detected in the right atrium (RA), the probe will be turned to the right side and the angle was adjusted to the ME bicaval view to confirm its entrance from the inferior vena cava. Then, the angle will be rapidly re-adjusted to view the ME right ventricle (RV) inflow-outflow view to confirm the extent of air embolism through the right ventricular outflow tract (RVOT).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea